CLINICAL TRIAL: NCT06204835
Title: ITGA6 Targeting NIR-II Fluorescence Image Guided Surgery of HCC Patients
Brief Title: ITGA6 Targeting NIR-II Fluorescence Image Guided Surgery
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Automation, Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Zhenhua Hu, Professor, Institute of Automation, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ITGARD7
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RDCy7 Intraoperative Fluorescence (Experimental): The patients will receive an injection of fluorophore (RDCy7) before the surgery. Then intraoperative fluorescence imaging will be performed to guide lesion resection.
  Interventions: Drug: RD-Cy7 fluorophore

INTERVENTIONS:
Drug: RD-Cy7 fluorophore — Fluorophore targeting ITGA6 that is overexpressed in HCC cells

SUMMARY:
In this study, the investigators will detect hepatocellular carcinoma lesions using fluoescence imaging with ITGA6 targeting probes during tumor resection surgery. The aim is to evaluate wether intraoperative fluorescence imaging targeting ITGA6 can help to improve the detction effect of hepatocellular carcinoma, and finally help the accurate surgical resection.

The main purposes of this study include:

1. To raise the detection rate of hepatocellular carcinoma intraoperatively using the novel NIR-II fluorescence molecular imaging and the ITGA6 targeting probe.
2. To validate the safety and effectiveness of the proposed ITGA6 targeting probes for clinical application.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been diagnosed with hepatocellular carcinoma.
2. Planned to receive hepatectomy.
3. Liver function Child-Pugh A.
4. ITGA6 was validated highly expressed preoperatively.
5. Aged 18 to 80, and the expected lifetime is longer than 6 months.
6. Approved to sign the informed consent.

Exclusion Criteria:

1. Allergic to Cy7.
2. Enrolled in other trials in the past 3 months.
3. Another malignant tumor was found.
4. Undesirable function of heart, lung, kidney, or any other organs.
5. Unable to tolerate a hepatectomy.
6. The researchers considered inappropriate to be included.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-07 (Actual); Primary Completion 2034-12-31 (Estimated); Study Completion 2039-12-31 (Estimated)

PRIMARY OUTCOMES:
HCC lesions | During hepatocellular resection surgery.
  Numbers of intraoperatively detected hepatocellular carcinoma lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenhua Hu, Ph. D, Principal Investigator — Institute of Automation, Chinese Academy of Sciences
Locations (2):
- China (2):
  - Guangdong, Guangzhou, Guangdong
  - Sichuan, Luzhou, Sichuan

IPD SHARING:
Plan to Share IPD: No
No publications available